CLINICAL TRIAL: NCT02590978
Title: Early Cholecystectomy in Patients With Mild Gallstone Acute Pancreatitis: A Randomized Prospective Study
Brief Title: Early Cholecystectomy in Patients With Mild Gallstone Acute Pancreatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis (n=52) with significantly differences in primary outcome (LOS)
Sponsor: Hospital del Salvador (Other)
Responsible Party: Principal Investigator, FRANCISCO RIQUELME, SURGEON, Hospital del Salvador
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPPAL-2015
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2015-12

CONDITIONS: Gallstone Pancreatitis
Keywords: gallstone pancreatitis; mild acute pancreatitis; adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early cholecystectomy (Experimental): Cholecystectomy within the first 72 hours of admission.
  Interventions: Procedure: Early cholecystectomy
- Control (Delayed cholecystectomy) (Other): Standard care arm. Cholecystectomy is delayed until normalization of laboratory values, abdominal pain resolves and oral intake is restored.
  Interventions: Procedure: Control (Delayed cholecystectomy)

INTERVENTIONS:
Procedure: Early cholecystectomy — Cholecystectomy + intraoperative cholangiography within the first 72 hours of admission.
  Arms: Early cholecystectomy
Procedure: Control (Delayed cholecystectomy) — Standard care arm. Cholecystectomy + intraoperative cholangiography is delayed once complete resolution of abdominal tenderness, oral feeding and trending down in pancreatic laboratory is achieved
  Arms: Control (Delayed cholecystectomy)

SUMMARY:
Randomized controlled trial to demonstrate the safety of early cholecystectomy (<72h) in patients with mild gallstone pancreatitis. The purpose of this study is to demonstrate that there is a shorter hospital stay and no higher complication rates.

DETAILED DESCRIPTION:
Acute pancreatitis is a prevalent disease, responsible for 220.000 hospital admissions per year in the United States of America. In Chile, during year 2012 there were 76.463 hospital admissions for this diagnosis, with a mean hospital stay of 11,8 days and 25 deaths per year associated with this disease (250 deaths from 2002 to 2012). The most frequent etiology of pancreatitis in Chile is gallstones, which can be present in 80% of the patients admitted for acute pancreatitis. This can be explained by the high prevalence of gallstones among these patients.

Since Acosta and Ledesma demonstrated the association between gallstones and acute pancreatitis in 1974, cholecystectomy has been the most efficient treatment option to prevent recurrence that can reach even 30-40% in the first two weeks after the first episode. There is consensus in delaying the time of the cholecystectomy in patients with acute gallstone pancreatitis where mortality can be as high as 80% in patients presenting with severe cases. However, the vast majority of the patients will present with a mild pancreatitis requiring no more than basic medical support. In these patients, the role of surgery during the same hospital admission has been clearly demonstrated.

There is no current consensus with respect to the safety of performing cholecystectomy in patients with mild pancreatitis within 48 to 72 hours after the hospital admission. There are few well-designed observational studies and only one randomized clinical trial, which has demonstrated a significant decrease in hospital stay (7 to 4 days), without increasing the rate of complications or mortality. According to some models of analysis and decision, this strategy could reduce costs associated with prolonged hospital stays and improve the quality of life of these patients without jeopardizing patient safety.

ELIGIBILITY:
Patients aged 18-70 years admitted with first gallstone acute pancreatitis (GAP) is evaluated for eligibility. Diagnosis and severity of GAP is based upon Atlanta Consensus modified at 2012. Acute pancreatitis is diagnosed when at least two out of three criteria are met; acute upper abdominal pain, elevated serum amylase/lipase level (more than thrice upper limit of normal range) and evidence of pancreatitis at any imaging modality (abdominal ultrasonography, computed tomography or magnetic resonance image). Biliary etiology is verified by abdominal ultrasonography showing stones or sludge at gallbladder. All other etiologies should be excluded. Exclusions criteria: (1) acute cholecystitis at abdominal ultrasonography, (2) suspected or confirmed acute cholangitis according to 2013 Tokyo Guidelines (fever or laboratory data with inflammatory response, cholestasis and imaging study with biliary dilatation/evident etiology), (3) history of Roux en Y gastric by pass or open supraumbilical surgery, (4) acute alcohol consumption, (5) chronic hepatic/pancreatic disease, (6) comorbidities contraindicating emergency surgery, (7) mental condition that preclude informed consent, (8) pregnancy, (9) patient refusal, (10) no endoscopist availability. There is no exclusions based on choledocolithiasis risk. All patients must complete clinical, anthropometric, and general laboratory/liver function tests at admission and daily until third day of stay or surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Length of Stay (LOS) | 90 dias
  days

SECONDARY OUTCOMES:
Endoscopic retrograde cholangio-pancreatography (ERCP) | 90 days
  yes/no
Conversion | surgery
  yes/no
Wound infection | 30 days
  yes/no
Re-admission | 90 days
  yes/no
Biliary complications | 90 days
  biloma, bile leak, residual choledocholithiasis
Operative time | surgery
  operative time in minutes
medical complications | 30 days
  any medical complication using Clavien-dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Riquelme, M.D., Principal Investigator — Universidad de Chile- Hospital del Salvador
Locations (1):
- Boris Marinkovic, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Ito K, Ito H, Whang EE. Timing of cholecystectomy for biliary pancreatitis: do the data support current guidelines? J Gastrointest Surg. 2008 Dec;12(12):2164-70. doi: 10.1007/s11605-008-0603-y. Epub 2008 Jul 18. PMID 18636298
- [Background] Kelly TR, Wagner DS. Gallstone pancreatitis: a prospective randomized trial of the timing of surgery. Surgery. 1988 Oct;104(4):600-5. PMID 3175860
- [Background] van Baal MC, Besselink MG, Bakker OJ, van Santvoort HC, Schaapherder AF, Nieuwenhuijs VB, Gooszen HG, van Ramshorst B, Boerma D; Dutch Pancreatitis Study Group. Timing of cholecystectomy after mild biliary pancreatitis: a systematic review. Ann Surg. 2012 May;255(5):860-6. doi: 10.1097/SLA.0b013e3182507646. PMID 22470079
- [Background] Cameron DR, Goodman AJ. Delayed cholecystectomy for gallstone pancreatitis: re-admissions and outcomes. Ann R Coll Surg Engl. 2004 Sep;86(5):358-62. doi: 10.1308/147870804227. PMID 15333174
- [Background] Aboulian A, Chan T, Yaghoubian A, Kaji AH, Putnam B, Neville A, Stabile BE, de Virgilio C. Early cholecystectomy safely decreases hospital stay in patients with mild gallstone pancreatitis: a randomized prospective study. Ann Surg. 2010 Apr;251(4):615-9. doi: 10.1097/SLA.0b013e3181c38f1f. PMID 20101174
- [Background] Randial Perez LJ, Fernando Parra J, Aldana Dimas G. [The safety of early laparoscopic cholecystectomy (<48 hours) for patients with mild gallstone pancreatitis: a systematic review of the literature and meta-analysis]. Cir Esp. 2014 Feb;92(2):107-13. doi: 10.1016/j.ciresp.2013.01.024. Epub 2013 Oct 4. Spanish. PMID 24099593
- [Background] Gurusamy KS, Nagendran M, Davidson BR. Early versus delayed laparoscopic cholecystectomy for acute gallstone pancreatitis. Cochrane Database Syst Rev. 2013 Sep 2;2013(9):CD010326. doi: 10.1002/14651858.CD010326.pub2. PMID 23996398
- [Background] Morris S, Gurusamy KS, Patel N, Davidson BR. Cost-effectiveness of early laparoscopic cholecystectomy for mild acute gallstone pancreatitis. Br J Surg. 2014 Jun;101(7):828-35. doi: 10.1002/bjs.9501. Epub 2014 Apr 23. PMID 24756933
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Derived] Riquelme F, Marinkovic B, Salazar M, Martinez W, Catan F, Uribe-Echevarria S, Puelma F, Munoz J, Canals A, Astudillo C, Uribe M. Early laparoscopic cholecystectomy reduces hospital stay in mild gallstone pancreatitis. A randomized controlled trial. HPB (Oxford). 2020 Jan;22(1):26-33. doi: 10.1016/j.hpb.2019.05.013. Epub 2019 Jun 22. PMID 31235428
- See also: Ministry of Public Health of Chile — http://www.minsal.cl/